CLINICAL TRIAL: NCT02309411
Title: 30-day, Single-arm Study of the Safety, Efficacy and the Pharmacokinetic and Pharmacodynamic Properties of Oral Rivaroxaban in Young Children With Various Manifestations of Venous Thrombosis
Brief Title: EINSTEIN Junior Phase II: Oral Rivaroxaban in Young Children With Venous Thrombosis
Acronym: EINSTEINJr
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14374; 2014-000566-22 (EudraCT Number)
Record Dates: First submitted 2014-11-24; First posted 2014-12-05 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Venous Thromboembolism
Keywords: Pediatric
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rivaroxaban (Experimental): Age and body weight-adjusted twice daily dosing of rivaroxaban to achieve a similar exposure as that observed in adults treated for venous thromboembolism (VTE) with 20 mg rivaroxaban once daily
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — With age and body-weight adjusted twice daily dosing of rivaroxaban as Oral Suspension to achieve a similar exposure as that observed in adults treated with 20 mg rivaroxaban once daily, and no other anticoagulant

SUMMARY:
The purpose of this study is to find out whether rivaroxaban is safe to use in children and how long it stays in the body. Safety will be assessed by looking at the incidence and types of bleeding events. There will also be a check for worsening of blood clots.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to < 6 years who have been treated for at least 2 months or, in case of catheter related thrombosis, for at least 6 weeks with LMWH (low molecular weight heparin), fondaparinux and/or VKA (vitamin K antagonist) for documented symptomatic or asymptomatic venous thrombosis - Hemoglobin, platelets, creatinine, alanine aminotransferase (ALT) and bilirubin evaluated within 10 days prior to randomization
* Informed consent provided

Exclusion Criteria:

* Active bleeding or high risk for bleeding contraindicating anticoagulant therapy
* Symptomatic progression of venous thrombosis during preceding anticoagulant treatment
* Planned invasive procedures, including lumbar puncture and removal of non peripherally placed central lines during study treatment
* An estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2
* Hepatic disease which is associated with either: coagulopathy leading to a clinically relevant bleeding risk, or ALT> 5x upper level of normal (ULN) or total bilirubin > 2x ULN with direct bilirubin > 20% of the total
* Platelet count < 50 x 10*9/L
* Hypertension defined as > 95th age percentile
* Life expectancy < 3 months
* Concomitant use of strong inhibitors of both cytochrome P450 isoenzyme 3A4 (CYP3A4) and P-glycoprotein (P-gp), i.e. all human immunodeficiency virus protease inhibitors and the following azole antimycotics agents: ketoconazole, itraconazole, voriconazole, posaconazole, if used systemically
* Concomitant use of strong inducers of CYP3A4, i.e. rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine
* Hypersensitivity or any other contraindication listed in the local labeling for the comparator treatment or experimental treatment
* Inability to cooperate with the study procedures
* Previous randomization to this study
* Participation in a study with an investigational drug or medical device within 30 days prior to randomization

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- United States (5):
  - Gainesville, Florida
  - Pensacola, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
- Parkville, Victoria, Australia
- Vienna, Austria
- Brazil (2):
  - São Paulo, São Paulo
  - São Paulo
- Toronto, Ontario, Canada
- Budapest, Hungary
- Israel (2):
  - Jerusalem
  - Ramat Gan
- Italy (3):
  - Milan, Lombardy
  - Turin, Piedmont
  - Padua, Veneto
- Setagaya City, Tokyo, Japan
- Nijmegen, Netherlands
- Poland (2):
  - Gdansk
  - Olsztyn
- Russia (3):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
- Spain (2):
  - Barcelona
  - Valencia
- Bern, Switzerland
- United Kingdom (3):
  - Newcastle upon Tyne, Tyne and Wear
  - Birmingham, West Midlands
  - Cardiff

REFERENCES:
- [Derived] Monagle P, Lensing AWA, Thelen K, Martinelli I, Male C, Santamaria A, Samochatova E, Kumar R, Holzhauer S, Saracco P, Simioni P, Robertson J, Grangl G, Halton J, Connor P, Young G, Molinari AC, Nowak-Gottl U, Kenet G, Kapsa S, Willmann S, Pap AF, Becka M, Twomey T, Beyer-Westendorf J, Prins MH, Kubitza D; EINSTEIN-Jr Phase 2 Investigators. Bodyweight-adjusted rivaroxaban for children with venous thromboembolism (EINSTEIN-Jr): results from three multicentre, single-arm, phase 2 studies. Lancet Haematol. 2019 Oct;6(10):e500-e509. doi: 10.1016/S2352-3026(19)30161-9. Epub 2019 Aug 13. PMID 31420317
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 27 study centers in 14 countries: Australia, Austria, Brazil, Canada, Hungary, Israel, Italy, Japan, Netherlands, Russia, Spain, Switzerland, United Kingdom, and United States between 15 January 2015 (first subject first visit) and 05 April 2017 (last subject last visit).
Pre-assignment Details: Overall, 51 subjects were screened, of these 5 subjects were screen failures; 4 subjects withdrew from study and 1 subject failed screening. Total of 46 subjects were assigned to treatment with 6 subjects received anticoagulant comparator (standard of care) and 40 subjects received rivaroxaban.
Groups:
- Rivaroxaban, Suspension, BID, Age: 2-6 Years: Subjects aged from 2 to 6 years were administered with age- and body weight-adjusted dose of rivaroxaban (BAY59-7939) oral suspension twice daily (BID) under fed conditions for 30 days.
- Rivaroxaban Suspension, BID, Age: 6 Months-2 Years: Subjects aged from 6 months to 2 years were administered with age- and body weight-adjusted dose of rivaroxaban oral suspension BID under fed conditions for 30 days.
- Anticoagulants, Comparator, Age: 2-6 Years: Subjects aged from 2 to 6 years were received comparator as per standard of care.
Period: Overall Study
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years | Anticoagulants, Comparator, Age: 2-6 Years
Started | 25 | 15 | 6
Completed | 23 | 14 | 6
Not Completed | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years | Anticoagulants, Comparator, Age: 2-6 Years | Total
Number analyzed (Participants) | 25 | 15 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.77 (1.03) | 1.26 (0.45) | 3.67 (0.82) | 2.94 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 3 | 24
  Male | 13 | 6 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 23 | 10 | 6 | 39
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Major Bleeding and Clinically Relevant Non-Major Bleeding Events
Description: Major bleeding is defined as overt bleeding and:
  * associated with a fall in hemoglobin of 2 gram/decilitre (g/dL) or more, or
  * leading to a transfusion of the equivalent of 2 or more units of packed red blood cells or whole blood in adults, or
  * occurring in a critical site, for example (e.g.) intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal, or
  * contributing to death.
  Clinically relevant non-major bleeding is defined as overt bleeding not meeting the criteria for major bleeding, but associated with:
  * medical intervention, or
  * unscheduled contact (visit or telephone call) with a physician, or
  * cessation (temporary) of study treatment, or
  * discomfort for the child such as pain or
  * impairment of activities of daily life (such as loss of school days or hospitalization).
Time Frame: During or within 2 days after stop of study treatment (up to 32 days)
Population: SAF included all subjects who received at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 25 | 15
Participants
  Major bleeding events | 0 | 0
  Clinically relevant non-major bleeding events | 0 | 0

2. Secondary Outcome: Number of Subjects With Symptomatic Recurrent Venous Thromboembolism
Description: Venous thromboembolism is the formation of a blood clot (thrombus) inside a blood vessel, obstructing the flow of blood through the circulatory system. The occurrence of recurrent venous thromboembolism was summarized by age group. Symptomatic recurrence, which is the composite of deep Vein Thrombosis (DVT), non-fatal Pulmonary Embolism (PE), and fatal PE of venous thrombosis, had to be documented using appropriate (repeat) imaging test.
Time Frame: From start of the study treatment up to 30-days post study treatment period (approximately 60 days)
Population: FAS included all enrolled children (before Amendment 4, all children were randomized by interactive voice/web response system [IxRS], after Amendment 4 all children were assigned to rivaroxaban by IxRS). Screening failures were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 25 | 15
Participants | 0 | 0

3. Secondary Outcome: Number of Subjects With Asymptomatic Deterioration in Thrombotic Burden on Repeat Imaging
Description: The occurrence of asymptomatic deterioration in thrombotic burden was summarized by age group. At the end of the 30-day treatment period, a repeat imaging of the thrombus was performed. The images of the index event and repeat imaging were adjudicated by the central independent adjudication committee (CIAC). The thrombotic burden at the time of the index event was compared to the thrombotic burden at the time of repeat imaging. The outcome of the adjudication was classified as normalized, improved, no relevant change, deteriorated, or not evaluable. Due to missing repeated imaging, thrombotic burden assessments were not done in some subjects.
Time Frame: At the end of the 30-day treatment period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 25 | 15
Participants
  Normalized | 6 | 4
  Improved | 15 | 4
  No relevant change | 1 | 3
  Deteriorated | 0 | 0
  Not evaluable | 0 | 0
  Not available | 0 | 0
  Missing | 3 | 4

4. Secondary Outcome: Change From Baseline in Prothrombin Time at Specified Time Points
Description: Prothrombin time is a global clotting test used for the assessment of the extrinsic pathway of the blood coagulation cascade. Day 30 (10-16 hours post-dose) was considered as a baseline.
Time Frame: Day 1 (2.5-4 hours post-dose); Day 15 (2-8 hours post-dose); Day 30 (10-16 hours post-dose)
Population: PDS with evaluable subjects for this end point. PD parameters were evaluated only for subjects who received active study medication.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 22 | 14
Seconds
  Day 1: 2.5-4 hours post-dose | 2.777 (4.845) | 2.514 (3.53)
  Day 15: 2-8 hours post-dose | 2.586 (2.387) | 4.764 (4.738)

5. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time at Specified Time Points
Description: The Activated partial thromboplastin time (aPTT) is a screening test for the intrinsic pathway. Day 30 (10-16 hours post-dose) was considered as a baseline.
Time Frame: Day 1 (2.5-4 hours post-dose); Day 15 (2-8 hours post-dose); Day 30 (10-16 hours post-dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 22 | 14
Seconds
  Day 1: 2.5-4 hours post-dose | 6.455 (17.036) | -3.479 (40.443)
  Day 15: 2-8 hours post-dose | 2.814 (6.375) | 21 (66.761)

6. Secondary Outcome: Concentration of Rivaroxaban in Plasma as a Measure of Pharmacokinetics at Specified Time Points
Description: Concentration of rivaroxaban in plasma was measured at Day 1, 15 and 30 at specified time points. In the below table, 'n' signifies those subjects who were evaluable for this measure at given time points for each group. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Day 1 (30-90 minutes, 2.5-4 hours post-dose); Day 15 (2-8 hours post-dose) and Day 30 (10-16 hours post-dose)
Population: PKS included all subjects with at least one pharmacokinetic sample in accordance with the pharmacokinetic sampling strategy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 24 | 15
microgram per liter (mcg/L)
  Day 1: 30-90 minutes post-dose | 72.8494 (153.76) | 68.0072 (160.77)
  Day 1: 2.5-4 hours post-dose: number analyzed (Participants) | 24 | 14
  Day 1: 2.5-4 hours post-dose | 108.6053 (58.18) | 76.5371 (112.91)
  Day 15: 2-8 hours post-dose: number analyzed (Participants) | 24 | 14
  Day 15: 2-8 hours post-dose | 112.3578 (46.37) | 61.3817 (451.46)
  Day 30: 10-16 hours post-dose: number analyzed (Participants) | 23 | 14
  Day 30: 10-16 hours post-dose | 19.8714 (189.49) | 5.9545 (354.51)

7. Other Pre Specified Outcome: Anti-factor Xa Values at Specified Time Points
Description: The individual anti-Factor Xa activity was determined ex-vivo using a photometric method. The anti-factor Xa assay is designed to measure plasma heparin, low molecular weight heparin and other anticoagulants. In the below table, 'n' signifies those subjects who were evaluable for this measure at given time points for each group.
Time Frame: Day 1 (2.5-4 hours post-dose); Day 15 (2-8 hours post-dose) and Day 30 (10-16 hours post-dose)
Population: PDS included all subjects with at least one blood sample for clotting tests in accordance with the pharmacodynamic sampling strategy was included.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban, Suspension, BID, Age: 2-6 Years | Rivaroxaban Suspension, BID, Age: 6 Months-2 Years
Number analyzed (Participants) | 22 | 14
microgram per liter (mcg/L)
  Day 1: 2.5-4 hours post-dose | 128.457 (69.615) | 87.831 (84.178)
  Day 15: 2-8 hours post-dose: number analyzed (Participants) | 22 | 13
  Day 15: 2-8 hours post-dose | 103.105 (58.343) | 131.369 (96.489)
  Day 30: 10-16 hours post-dose | 19.069 (17.463) | 16.952 (19.725)

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 day post study treatment (approximately 60 days)
Groups:
- Rivaroxaban BID (Suspension) (2 - 6 Years Group): Subjects aged from 2 to 6 years were administered with age- and body weight-adjusted dose of rivaroxaban oral suspension BID under fed conditions for 30 days.
- Rivaroxaban BID (Suspension) (6 Months - 2 Years Group): Subjects aged from 6 months to 2 years were administered with age- and body weight-adjusted dose of rivaroxaban oral suspension BID under fed conditions for 30 days.
- Anticoagulants, Comparator (2 - 6 Years Group): Subjects aged from 2 to 6 years were received comparator as per standard of care.
Arm/Group | Rivaroxaban BID (Suspension) (2 - 6 Years Group) | Rivaroxaban BID (Suspension) (6 Months - 2 Years Group) | Anticoagulants, Comparator (2 - 6 Years Group)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/25 | 2/15 | 1/6
Other Adverse Events (participants affected / at risk) | 14/25 | 11/15 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban BID (Suspension) (2 - 6 Years Group) (N=25) | Rivaroxaban BID (Suspension) (6 Months - 2 Years Group) (N=15) | Anticoagulants, Comparator (2 - 6 Years Group) (N=6)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban BID (Suspension) (2 - 6 Years Group) (N=25) | Rivaroxaban BID (Suspension) (6 Months - 2 Years Group) (N=15) | Anticoagulants, Comparator (2 - 6 Years Group) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal erosion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 1 (2) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bronchoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study started as randomized but the Comparator arm sample size was too small for meaningful comparison; it was removed in Protocol amendment and approved by review board. Results only reported for rivaroxaban arm as single arm study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02309411/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02309411/SAP_001.pdf